CLINICAL TRIAL: NCT01718301
Title: A Study to Evaluate Safety and Efficacy of Boceprevir-response Guided Therapy in Controlled HIV Patients With Chronic Hepatitis C Genotype 1 Infection Who Failed Previously to Peginterferon /Ribavirin Eudra CT2012-003984-23
Brief Title: HIV Patients With Chronic Hepatitis C Genotype 1 Infection Who Failed Previously to Peginterferon /Ribavirin
Acronym: BOC-HIV
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty in patient recruitment
Sponsor: Anna Cruceta (Other)
Responsible Party: Sponsor-Investigator, Anna Cruceta, Clinical Research manager, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BOC-HIV; 2012-003984-23 (EudraCT Number)
Record Dates: First submitted 2012-10-25; First posted 2012-10-31 (Estimated); Results first posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Hepatitis C; HIV Infections; COINFECTION
Keywords: HCV; HIV; Coinfection
MeSH Terms: conditions — Hepatitis C; HIV Infections; Coinfection | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; Ribavirin; peginterferon alfa-2a; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- boceprevir + ribavirin + peginterferon (Experimental): boceprevir 800 mg three times a day (v.o.) in combination with peginterferon (alfa-2b or alfa-2a) and ribavirin
  Interventions: Drug: boceprevir; Drug: Ribavirin; Drug: Peginterferon alfa-2a; Drug: Peginterferon alfa-2b

INTERVENTIONS:
Drug: boceprevir
Drug: Ribavirin
Drug: Peginterferon alfa-2a
Drug: Peginterferon alfa-2b

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of a Response Guided Therapy of boceprevir 800 mg dosed three times a day (TID) orally (PO) in combination with Peginterferon (either alpha 2b or alpha 2a) and Ribavirin in HIV/HCV genotype 1 infected patients that failed to previous HCV therapy.

DETAILED DESCRIPTION:
In a total number of 108 patients the protocol was evaluated but only in 102 the protocol efectively was presented. In the remaining 6 patients we don't believe the trial could be performed.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion in the study, subjects must have a qualifying regimen defined as peginterferon alfa-2a plus ribavirin or peginterferon alfa-2b plus ribavirin for a minimum of 12 weeks. If a subject has received more than one such regimen, the most recent regimen is considered the qualifying regimen.
* Subject must have previously documented chronic hepatitis C (CHC) genotype 1 infection. Subjects with other or mixed genotypes are not eligible. The HCV-RNA result at the screening visit must confirm genotype 1 infection and be ≥10,000 IU/mL.
* Subject must have a liver biopsy with histology consistent with CHC and no other etiology and/or Fibroscan assessment. In case of:

  1. No cirrhosis. Biopsies and/or Fibroscan must be within 18 months of screening visit.
  2. Cirrhosis. No specific length of time would be requested.
* All patients with cirrhosis must have an ultrasound 6 month within of screening visit.
* Patients must be on stable antiretroviral therapy including a CD4 cell count of more than 100 per mm3 and a HIV plasmatic viral load undetectable (it is < 50 copies/mL) for more than 6 months. Antiretroviral therapy must be Raltegravir-based (al least during the last 3 months).
* Subject must be ≥18 years of age.
* HIV treatment should not contain efavirenz (EFV), nevirapine (NVP), etravirine (ETV), didanosine (ddI), stavudine (d4T), zidovudine (AZT), or HIV protease inhibitors.
* Subject must weight between 40 kg and 125 kg.
* Subject and subject's partner(s) must each agree to use acceptable methods of contraception for at least 2 weeks prior to Day 1 and continue until at least 6 months after last dose of study drug.
* Subjects must be willing to give written informed consent and by investigator opinion be able to follow the protocol visit design.

Exclusion Criteria:

* Subjects known to be coinfected with hepatitis B virus (HBsAg positive).
* Patients chronically infected with HCV genotype other than 1
* CD4 cell count < 100 cel/mm3.
* Plasma HIV RNA more than 50 copies/mL
* Platelet count less than 80.000 /mm3
* Subjects who required discontinuation of previous interferon or ribavirin regimen for a severe adverse event considered by the investigator to be possibly or probably related to ribavirin and/or interferon.
* Treatment with ribavirin within 90 days and any interferon-alpha within 1 month of Screening.
* Treatment for hepatitis C with any investigational medication. Prior treatments with herbal remedies with known hepatotoxicity are exclusionary.
* Participation in any other clinical trial within 30 days of randomization or intention to participate in another clinical trial during participation in this study.
* History of hemoglobinopathy (e.g., thalassemia) or any other cause of or tendency to hemolysis.
* Evidence of decompensate liver disease including, but not limited to, a history or presence of clinical ascites, bleeding varices, or hepatic encephalopathy.
* Diabetic and/or hypertensive subjects with clinically significant ocular examination findings.
* Unstable or untreated pre-existing psychiatric condition.
* Any known pre-existing medical condition that could interfere with the subject's participation in and completion of the study.
* Any current evidence of substance abuse of alcohol or other drugs.
* Subjects receiving opioid agonist substitution therapy but not enrolled in an opiate substitution maintenance program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2013-03-10 (Actual); Primary Completion 2015-03-20 (Actual); Study Completion 2015-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josep Mallolas, MD, Principal Investigator — Hospital Clínic i Provincial de Barcelona
Locations (1):
- Hospital Clinic i Provincial de Barcelona, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Started 21/06/2013 and finished 04/12/2013
Groups:
- Boceprevir + Ribavirin + Peginterferon: Participants received 4 weeks of Peginterferon/Ribavirin (lead-in), followed by response-guided therapy with Boceprevir added. Cirrhotic patients received a fixed 44-week regimen.
  Boceprevir 800 mg three times a day (v.o.) in combination with Peginterferon (alfa-2b or alfa-2a) and Ribavirin
Period: Overall Study
Arm/Group | Boceprevir + Ribavirin + Peginterferon
Started | 102 (Study started on 21/06/2013)
Completed | 98 (Study was finished on April 2015)
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- Boceprevir Plus Peginterferon/Ribavirin to Retreat HCV Genotyp: boceprevir 800 mg three times a day (v.o.) in combination with peginterferon (alfa-2b or alfa-2a) and ribavirin
Arm/Group | Boceprevir Plus Peginterferon/Ribavirin to Retreat HCV Genotyp
Number analyzed (Participants) | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 73
Region of Enrollment [Number; unit: participants]
  Spain | 98

OUTCOME MEASURES:

1. Primary Outcome: Achievement of Sustained Virological Response (SVR) at 24 Weeks Post-Treatment
Description: Achievement of SVR, defined as undetectable plasma HCV-RNA at Follow-up Week (FW) 24.
  If a subject is missing FW 24 data and has undetectable HCV-RNA level at FW 12, the subject would be considered an SVR.
Time Frame: Week 24
Population: All patients who received at least one dose of study medication were included in the efficacy analysis.
  Patients with detectable HCV RNA at week 12 were discontinued per protocol-defined futility criteria.
Measure: Count of Participants; unit: Participants
Groups:
- Boceprevir + Ribavirin + Peginterferon: boceprevir 800 mg three times a day (v.o.) in combination with peginterferon (alfa-2b or alfa-2a) and ribavirin
  boceprevir
  Ribavirin
  Peginterferon alfa-2a
  Peginterferon alfa-2b
Arm/Group | Boceprevir + Ribavirin + Peginterferon
Number analyzed (Participants) | 98
Participants
  Number of participants achieving SVR | 66
  Number of participants not achieving SVR | 32

2. Secondary Outcome: Achievement of Sustained Virological Response at Weeks 2,4,8,12.
Description: Proportion of participants with undetectable HCV RNA (<15 IU/mL) at weeks 2, 4, 8, and 12 during treatment.
Time Frame: Weeks 2, 4, 8, 12
Reporting Status: Not Posted

3. Secondary Outcome: The Proportion of Subjects With Undetectable HCV-RNA at FW 12.
Description: The proportion of subjects with undetectable HCV-RNA at follow-up week 12.
Time Frame: Week 12
Reporting Status: Not Posted

4. Secondary Outcome: The Proportion of Subjects With Undetectable HCV-RNA at 72 Weeks After Randomization.
Description: The proportion of randomized subjects with undetectable HCV-RNA at 72 weeks after randomization.
Time Frame: Week 72
Reporting Status: Not Posted

5. Secondary Outcome: Number of Adverse Events
Description: Safety: number of adverse events
Time Frame: From baseline to study completion (up to 72 weeks)
Reporting Status: Not Posted

6. Secondary Outcome: Resistance of HCV After Boceprevir (BOC) Containing Regimen
Description: Resistance of HCV after boceprevir containing regimen. Blood samples will be collected at baseline and after HCV virological failure and resistance analysis will be done at the end of the study in a single Center (Hospital Clínic-Barcelona).
Time Frame: whenever resistance occurs during the study (from week 12 until the date the resistance occurs, assessed up to 72 weeks)
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Boceprevir + Ribavirin + Peginterferon: Side effects leading to drug discontinuation appeared in 6 patients.
Arm/Group | Boceprevir + Ribavirin + Peginterferon
Serious Adverse Events (participants affected / at risk) | 6/98
Other Adverse Events (participants affected / at risk) | 1/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boceprevir + Ribavirin + Peginterferon (N=98)
Anemia (Blood and lymphatic system disorders) | 6 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boceprevir + Ribavirin + Peginterferon (N=98)
Headache (Psychiatric disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-09-18): https://cdn.clinicaltrials.gov/large-docs/01/NCT01718301/Prot_SAP_000.pdf